CLINICAL TRIAL: NCT06964490
Title: Effect of Different Apex Locators on Postoperative Pain in Endodontic Retreatment of Single-Rooted Teeth: Prospective Randomized Clinical Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ipek Eraslan Akyuz (Other)
Responsible Party: Sponsor-Investigator, Ipek Eraslan Akyuz, dentist, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/3
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Retreatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ProPex Pixi Apex Locator (Experimental)
  Interventions: Device: determination of working length
- Root ZX Apex Locator (Experimental)
  Interventions: Device: determination of working length
- Raypex 6 Apex Locator (Experimental)
  Interventions: Device: determination of working length

INTERVENTIONS:
Device: determination of working length — Compare the effect of WL determination using different apex locator devices (ProPex Pixi, Root ZX, and Raypex 6) on the incidence and intensity of postoperative pain following endodontic retreatment in single-rooted teeth

SUMMARY:
Nonsurgical endodontic retreatment is a vital procedure that promotes periapical healing by eliminating previous root canal fillings, necrotic tissue, and residual microorganisms, thanks to the comprehensive cleaning of the root canal system [1]. The successful disinfection of intricate anatomical structures, such as dentinal tubules, lateral canals, and isthmuses, largely depends on the effective removal of obturation materials [2]. Even in the absence of coronal leakage or recurrent caries, persistent clinical symptoms or radiographic evidence of periapical pathology may indicate treatment failure, warranting retreatment [3]. Residual bacteria and remnants of root filling materials are known contributors to posttreatment disease [4].

A key factor in the success of both primary endodontic treatment and retreatment is the accurate determination of working length (WL), which dictates the apical extent of canal instrumentation and obturation [5]. Inadequate WL may result in over-instrumentation, leading to periapical irritation and postoperative pain [6]. WL is generally defined as the distance from a coronal reference point to the location where canal cleaning, shaping, and filling should ideally terminate, often coinciding with the apical constriction, and occasionally with the cementodentinal junction, where pulpal and periodontal tissues transition [5].

Although periapical radiographs are still commonly used for WL determination, they do not always provide definitive results due to certain limitations. Factors such as improper film placement, angular distortion, image magnification and distortion, patient exposure to ionizing radiation, and the superimposition of anatomical structures can compromise the accuracy of measurements [7]. As a result, electronic apex locators (EALs) have gained prominence as a dependable and objective tool for determining WL, offering real-time measurements less influenced by operator variability or anatomical distortions [6].

The initial generations of electronic apex locators (EALs) exhibited inconsistent readings and limited accuracy, particularly in the presence of irrigation solutions or tissue fluids. However, recent advancements have significantly enhanced the reliability and clinical performance of EALs. Modern EALs, such as the ProPex Pixi (Dentsply, Switzerland) and Root ZX (J. Morita, Japan) apex locators, utilize multiple-frequency impedance measurements to detect changes as the file approaches the minor apical foramen [8]. These devices are equipped with microprocessors that analyze real-time impedance variations, allowing for dynamic and accurate assessment of canal length during instrumentation. Thanks to these technological enhancements, contemporary EALs can precisely identify the apical constriction, even under challenging clinical conditions [9]. Recent studies have demonstrated that modern devices can achieve up to 90% accuracy in WL determination, making them indispensable tools in both primary and secondary endodontic procedures [9, 10]. Raypex (Raypex 6, VDW GmbH, Munich, Germany) is another widely used electronic apex locator (EAL). Aydın et al. [11] demonstrated that Raypex 6 showed success rates of 85% and 95% within ±0.5 mm and ±1 mm, respectively, in teeth with mature apices. Although apex locators function with the same principle, the areas detected by different devices may differ. These variations in apical measurements among different EALs may not only affect treatment accuracy but could also influence the extent of postoperative pain experienced by the patient.

Postoperative pain is a significant concern in endodontics, with its incidence ranging from 3% to 58% [12]. Irritation of periradicular tissues during root canal treatment induces an acute inflammatory response, leading to the release of chemical mediators and changes in local pressure and tissue adaptation [13]. Accurate WL determination plays a critical role in minimizing postoperative pain [14]. Although the use of electronic EALs in WL determination during root canal treatment has been widely accepted, there are only a limited number of clinical studies investigating their effect on postoperative pain. Recent studies have explored the clinical performance and accuracy of different EALs; however, their focus was primarily on measurement precision rather than postoperative outcomes like pain or patient comfort [7, 15].

Despite the increasing use of EALs in endodontic procedures, there is currently no clinical study that examines the impact of using different apex locator devices on postoperative pain in the nonsurgical endodontic retreatment. Given the added complexity of retreatment cases, such as the need to remove previous obturation materials and the potential for greater periapical irritation, this represents a significant gap in the literature. The primary aim of this randomized clinical study is to evaluate and compare the effect of WL determination using different apex locator

ELIGIBILITY:
Inclusion Criteria:

* 1. ASA I or II individuals aged 18-60 years 2. Single-rooted, single-canaled teeth treated with root canal therapy ≥4 years ago 3. Root canal fillings ending 2-3 mm short of the radiographic apex 4. Diagnosis of asymptomatic apical periodontitis 5. Periapical Index (PAI) score of 2-4 [17], with no periodontal or prosthetic treatment needs 6. Root canal curvature <30° 7. Radiographically confirmed complete root formation and absence of resorption 8. Ability to achieve rubber dam isolation during treatment 9. Voluntary participation with signed informed consent

Exclusion Criteria:

* 1. Use of analgesics, antibiotics, or corticosteroids within the past two weeks 2. Periodontal attachment loss (probing depth > 4 mm) 3. Teeth with vertical root fractures, external resorption, or perforations 4. Teeth with fractured instruments inside the root canal system 5. Severe root curvature or excessive coronal destruction on preoperative radiographs 6. Canal calcification, root resorption, or incomplete root development 7. Cognitive impairment, mental retardation, or inability to comply due to old age 8. Pregnancy or lactation 9. Presence of systemic conditions (e.g., widespread infection, cancer, cardiovascular disease, advanced diabetes)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity Assessed by Visual Analog Scale (VAS) | From 6 hours up to 7 days after endodontic retreatment
  Postoperative pain intensity will be evaluated using the Visual Analog Scale (VAS), a 100-mm line where patients mark their pain level. VAS scores will be categorized as: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm). Patients will record their pain at 6, 12, and 24 hours postoperatively, and daily for up to 7 days following endodontic retreatment. Pain scores will be compared among the three apex locator groups (ProPex Pixi, Root ZX, Raypex 6) to assess the impact of different devices on postoperative pain levels.

IPD SHARING:
Plan to Share IPD: No